CLINICAL TRIAL: NCT04873960
Title: Translation of ECOS-16 Questionnaire in Urdu Language; Validity and Reliability Analysis in Postmenopausal Women With Osteopenia
Brief Title: Translation and Cross -Cultural Validation of ECOS-16 Questionnaire in Urdu Language
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/21/1102/A Saima Riaz
Record Dates: First submitted 2021-04-23; First posted 2021-05-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Postmenopausal Osteopenia; Quality of Life; Validity; Reliability; Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteopenia is a clinical term to define the declined Bone Mineral Density (BMD) as per the normal reference values but not low enough to meet osteoporotic diagnostic criteria. A Dual-energy x-ray absorptiometry (DXA) bone scan is used to diagnose decreased BMD. Osteopenia is, as described by the World Health Organization (WHO), a score ranging from -1 to -2.5, whereas Osteoporosis is diagnosed with values less than - 2.5. The risk of a decrease in BMD doubles as a woman goes into Menopause.

The objective of this study will be to determine the effects of Kinect-based virtual reality training on BMD, fracture risk, physical function and Quality of life in postmenopausal women with Osteopenia. The aim of the present study is to translate the ECOS-16 Questionnaire into Urdu Language along with validation of the translated versions by evaluating its validity and reliability in the Postmenopausal women of Pakistan with Osteopenia or Osteoporosis and understanding Urdu Language. No such study has been previously conducted in the Pakistan region which translates the specific questionnaire and follows the proper cross-culture adaptation protocol.

DETAILED DESCRIPTION:
ECOS-16 was developed to evaluate the quality of life in postmenopausal women with osteoporosis. It is a brief, straightforward, self-administered questionnaire containing 16 easy-to-score items, 4 of which are taken from OQLQ and the remaining 12 taken from the Questionnaire of the QUALEFFO-41 . The 16 items are further divided into four subscales: pain (5 items), physical functioning (5 items), illness-related fear (2 items), and psychosocial functioning (4 items). Each question related to these items has five response options, ranging from 1 to 5, where 5 represents the worst quality of life score. ECOS-16 provides both subscale domain scores and an overall score. ECOS-16 questionnaire, originally developed in English, has been translated into many languages to assess for its validity and reliability ever since, but Urdu version is not developed or tested. Previous studies have shown that the translation of the scale would end up giving a standard measure to be utilized in clinical practices and research studies while sanctioning clinicians and specialists to share information and have an insight into patient's health-related concerns of Osteoporosis. The reliability and validity of the ECOS-16 have been well documented by the developers of the instrument Thus, it is imperative to translate this questionnaire into psychometrically tested Urdu version. This may promote an easy understanding of the local population in Pakistan where the Urdu language is spoken and will provide a valid measure of Quality of life to be clinically utilized by practitioners and researchers across the country.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who can speak and understand the Urdu language
* Osteopenic with Lumbar spine or femur T-score between -1 to -2.5
* Osteoporotic with Lumbar spine or femur T-score less than -2.5.

Exclusion Criteria:

* Impairment of communicative and sensorial functions
* Impaired Cognition
* Unstable angina
* disease requiring oxygen therapy and Symptomatic orthostatic hypotension
* Hypertension in poor pharmacologic control (diastolic >95 mmHg, systolic >160 mmHg)
* Neurological disorders

Ages: 48 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women with Osteoporosis or Osteopenia
Study Population: Postmenopausal women diagnosed with Osteoporosis and Osteopenia , clinically stable, between age 48-70 years and able to read and complete the Urdu version of ECOS-16 Questionnaire. Women having any condition mentioned in exclusion criteria will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
ECOS-16 Quality of Life Questionnaire | 6 Months
  ECOS-16 evaluates the quality of life in postmenopausal women with osteoporosis. It is a brief, straightforward, self-administered questionnaire containing 16 easy-to-score items. The 16 items are further divided into four subscales: pain (5 items), physical functioning (5 items), illness-related fear (2 items), and psychosocial functioning (4 items). Each question related to these items has five response options, ranging from 1 to 5, where 5 represents the worst quality of life score. ECOS-16 provides both subscale domain scores and an overall score. Its translation is to be done in the local languages of Pakistan through a rigorous and approved process.

SECONDARY OUTCOMES:
Reliability of Urdu translated version | 6 Months
  To determine reliability of cross-culturally adapted and the Urdu translated version of ECOS-16 in postmenopausal women with Osteoporosis/Osteopenia. Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two or more intervals between different visits of the patient.
Validity of Urdu Translated version | 6 Months
  To determine validity of cross-culturally adapted and the Urdu translated version of ECOS-16 in postmenopausal women with Osteoporosis/Osteopenia. Validity is how accurate the tool measures an item it is supposed to. Thus these both are to be measured through various parameters to validate the translated version as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, PhD, Study Chair — Riphah International University; Saima Riaz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Saima Riaz, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badia X, Diez-Perez A, Lahoz R, Lizan L, Nogues X, Iborra J. The ECOS-16 questionnaire for the evaluation of health related quality of life in post-menopausal women with osteoporosis. Health Qual Life Outcomes. 2004 Aug 3;2:41. doi: 10.1186/1477-7525-2-41. PMID 15291959
- [Background] Salaffi F, Malavolta N, Cimmino MA, Di Matteo L, Scendoni P, Carotti M, Stancati A, Mule R, Frigato M, Gutierrez M, Grassi W; Italian Multicentre Osteoporotic Fracture (IMOF) Study Group. Validity and reliability of the Italian version of the ECOS-16 questionnaire in postmenopausal women with prevalent vertebral fractures due to osteoporosis. Clin Exp Rheumatol. 2007 May-Jun;25(3):390-403. PMID 17631735
- [Background] Abourazzak FE, Allali F, Rostom S, Hmamouchi I, Ichchou L, El Mansouri L, Bennani L, Khazzani H, Abouqal R, Hajjaj-Hassouni N. Factors influencing quality of life in Moroccan postmenopausal women with osteoporotic vertebral fracture assessed by ECOS 16 questionnaire. Health Qual Life Outcomes. 2009 Mar 13;7:23. doi: 10.1186/1477-7525-7-23. PMID 19284667
- [Background] Moradzadeh R, Moghimi N, Nadrian H, Behrouzi F, Keshavarz T, Golmohammadi P. Validity and reliability of the Farsi version of the ECOS-16 questionnaire for females with osteoporosis. East Mediterr Health J. 2018 Jan 2;23(11):729-733. doi: 10.26719/2017.23.11.729. PMID 29319144
- [Background] Lee JS, Son SM, Goh TS, Kim TH, Noh EY. Validation of the ECOS-16 Questionnaire in Koreans with Osteoporosis. Asian Spine J. 2016 Oct;10(5):877-885. doi: 10.4184/asj.2016.10.5.877. Epub 2016 Oct 17. PMID 27790315
- [Background] Madureira MM, Ciconelli RM, Pereira RM. Quality of life measurements in patients with osteoporosis and fractures. Clinics (Sao Paulo). 2012 Nov;67(11):1315-20. doi: 10.6061/clinics/2012(11)16. PMID 23184210